CLINICAL TRIAL: NCT01978496
Title: A Multicenter Double-blind, Randomized Placebo Controlled, Parallel Group, Study of the Efficacy and Safety of Oral Eletriptan in Subjects With Acute Migraine
Brief Title: Efficacy, Safety, and Tolerability of Oral Eletriptan for Treatment of Acute Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A160-102
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Migraine With or Without Aura
MeSH Terms: interventions — eletriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Eletriptan 20 mg (Experimental)
  Interventions: Drug: Eletriptan 20 mg
- Eletriptan 40 mg (Experimental)
  Interventions: Drug: Eletriptan 40 mg
- Eletriptan 80 mg (Experimental)
  Interventions: Drug: Eletriptan 80 mg

INTERVENTIONS:
Drug: Placebo — matching placebo
  Arms: Placebo
Drug: Eletriptan 20 mg — 20mg oral
  Arms: Eletriptan 20 mg
Drug: Eletriptan 40 mg — 40mg oral
  Arms: Eletriptan 40 mg
Drug: Eletriptan 80 mg — 80mg oral
  Arms: Eletriptan 80 mg

SUMMARY:
To confirm the efficacy of three dose levels of oral eletriptan relative to placebo in relieving symptoms of acute migraine and to further explore the dose response relationship of eletriptan.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one typical attack of migraine with or without aura every 6 weeks, as defined by the International Headache Society (IHS) criteria.
* Capable of taking study medication as outpatients and recording its effects.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Migraine subjects who also suffered from concomitant frequent (non-migraine) headache, defined as more than six headaches per month on average
* Migraine attacks that were thought to be atypical and had consistently failed to respond to medical therapy.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1334 (Actual)
Dates: Start 1996-07; Primary Completion 1997-12 (Actual); Study Completion 1997-12 (Actual)

PRIMARY OUTCOMES:
Headache responder rate at two hours after the first dose for the first attack. | 2 hours
  A headache response was defined as a subject having improvement in headache severity from grade 2 or 3 at baseline to 0 or 1 at two hours post-dose.

SECONDARY OUTCOMES:
Pain free responder rate at two hours after the first dose for the first attack. | 2 hours
  Pain free response was defined as improvement from grade 2 or 3 at baseline to grade 0 at two hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A160-102&StudyName=Efficacy%2C%20Safety%2C%20and%20Tolerability%20of%20Oral%20Eletriptan%20for%0ATreatment%20of%20Acute%20Migraine